CLINICAL TRIAL: NCT00006323
Title: Neurobehavioral Consequences of Sleep Apnea in Children
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 926; R01HL062371 (NIH)
Record Dates: First submitted 2000-10-02; First posted 2000-10-03 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-03

CONDITIONS: Lung Diseases; Sleep Apnea Syndromes
MeSH Terms: conditions — Lung Diseases; Sleep Apnea Syndromes

SUMMARY:
To identify physiological and clinical measures of obstructive sleep-disordered breathing that are associated with increased morbidity in children.

DETAILED DESCRIPTION:
BACKGROUND:

The study is in response to a Request for Applications (RFA) on Obstructive Sleep Apnea in Children. NHLBI issued the RFA in December, 1997, with co-sponsorship from the National Institute of Dental and Craniofacial Research and the National Institute of Child Health and Human Development.

DESIGN NARRATIVE:

This cross-sectional study recruited a population-based sample of young children from among the more than 8000 children in Massachusetts enrolled in the on-going Infant Care Practices Study. Stratified sampling was used to assemble a cohort of 250 children with habitual snoring (> 3 nights/week), 100 children with occasional snoring (<3 nights/week), and 100 non-snoring children. These children were studied within 3 months of their fourth birthday using overnight laboratory polysomnography and a detailed neurobehavioral evaluation, in order to test the hypothesis that, after adjusting for potential confounding variables, both parent-reported snoring and polysomnographic measures were associated with standardized measures of the following neurobehavioral domains: immediate attention, sustained attention, working memory, and symptoms of hyperactivity. These data also provided an opportunity to determine normal values for polysomnographic measures in 4-year-old children and to determine the prevalence of snoring and polysomnographic abnormalities among 4-year-old children.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-09; Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gottlieb — Boston University

REFERENCES:
- [Background] Gottlieb DJ, Vezina RM, Chase C, Lesko SM, Heeren TC, Weese-Mayer DE, Auerbach SH, Corwin MJ. Symptoms of sleep-disordered breathing in 5-year-old children are associated with sleepiness and problem behaviors. Pediatrics. 2003 Oct;112(4):870-7. doi: 10.1542/peds.112.4.870. PMID 14523179
- [Background] Gottlieb DJ, Chase C, Vezina RM, Heeren TC, Corwin MJ, Auerbach SH, Weese-Mayer DE, Lesko SM. Sleep-disordered breathing symptoms are associated with poorer cognitive function in 5-year-old children. J Pediatr. 2004 Oct;145(4):458-64. doi: 10.1016/j.jpeds.2004.05.039. PMID 15480367